CLINICAL TRIAL: NCT05570721
Title: The Comorbidity of Depression and Cardiovascular Disease in Midlife Women: Investigating Novel Biological Pathways of Risk
Brief Title: Depression, Aging, Stress and Heart Health Study
Acronym: DASHH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: The Foundation of Hope for Research and Treatment of Mental Illness (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 22-0763
Record Dates: First submitted 2022-09-27; First posted 2022-10-07 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Menopause; Depression; Heart Disease in Women; Stress
MeSH Terms: conditions — Depression | interventions — Psychological Tests

STUDY DESIGN:
Intervention Model Description: Participants will be exposed to a mental stress task (the TSST)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Women with perimenopausal depression (Experimental): Participants will undergo a social stress task (TSST)
  Interventions: Behavioral: Trier Social Stress Test
- Women without perimenopausal depression (Experimental): Participants will undergo a social stress task (TSST)
  Interventions: Behavioral: Trier Social Stress Test

INTERVENTIONS:
Behavioral: Trier Social Stress Test — The TSST has both social-evaluative and arithmetic components. During the social-evaluative component, the participant is asked to prepare and then deliver a brief speech to the research team. After this component there is a surprise arithmetic problem. This challenge paradigm has been well-established to rapidly and robustly induce psychological stress as well as physiological indices of stress (e.g., cortisol response, heart rate response). This task takes approximately 15 minutes to complete.

SUMMARY:
Depression is a known risk factor for cardiovascular disease (CVD), and this comorbidity contributes significantly to the morbidity and mortality of women. The menopausal transition or perimenopause is a period of vulnerability for both depression and CVD, making it a key time to study this critical public health issue. This research will preliminarily explore whether disruption in two novel stress pathways 1) the renin-angiotensin-aldosterone system (RAAS) and autonomic nervous system (ANS) and their relationship may underlie the link between these illnesses. Findings will provide important insight into potential mechanisms by which depression during perimenopause may increase risk for CVD in midlife women, which will inform potential risk reduction and treatment strategies that can improve health outcomes in this population.

DETAILED DESCRIPTION:
This study uses an experimental stress task to induce mild social stress and activation of two physiological stress pathways (the RAAS and ANS) that may be be involved in the association between perimenopausal depression and risk for cardiovascular disease in women. Perimenopausal women with mild-moderate depressive symptoms and healthy women without any psychiatric history will be enrolled. All participants will complete the same study procedures.

During the first visit (conducted remotely) consent will be obtained. After consent, participants will answer questions about their psychiatric history as part of a standardized psychological assessment (the Mini International Neuropsychiatric Interview) and medical/reproductive history, including current medications. They will also complete brief questionnaires about their current mood symptoms and history of exposure to trauma. Risk for self-harm using the Columbia Suicide Severity Rating Scale (CSSRS) will be assessed. After it is determined that a participant is eligible based on these assessments, she will then be given instruction for how to prepare for the second study visit, including refraining from exercise, alcohol, caffeine for at least 4 hours prior to the visit. Dietary education is also provided and participants are asked to keep a food journal for 3 days prior to the second study visit to standardize nutritional content prior to the second study visit.

During the second visit (conduced in-person in a laboratory setting) participants will complete a brief stress task. All of these visits will be conducted between 2-6 in the afternoon/evening.This visit will have four components:

1. Orientation: participants will be oriented to the study visit and taught how to do the saliva collection. Height and weight will be measured and a urine pregnancy test completed. The CSSRS will be repeated for safety.
2. Rest period: this includes a 30-minute resting period in the seated position. Participants will complete self-report questionnaires on mood, anxiety, sleep and menopausal symptoms. 2 electrocardiogram (EKG) leads and nodes will be applied for the heart rate monitoring portion. During any residual time white noise will be played and the lights dimmed to promote relaxation.
3. Completion of the stress task (the Trier Social Stress Test or TSST): this task involves social evaluation, speech, and math related stress and takes approximately 15 minutes to complete. Participants are introduced to a 1-2-person committee. The participant will assume the role of a job applicant who is invited for a personnel interview with the committee. Anticipation: The participant prepares for 5 minutes. Speech (5 mins): The committee asks the participant to deliver her talk for 5 minutes. The committee responds with prepared questions to ensure that the talk lasts for 5 minutes. Serial Subtraction (5 mins): The committee members will give the participant a number to start from and then ask them to subtract a number from that original number and then continue to subtract that same number, saying aloud the answers until they get to zero.
4. Recovery and debriefing: during this phase the participant rests alone. After recovery is complete the study team will debrief with the participant about the nature of stress task and answer any questions.

Sample collection: blood and saliva will be collected immediately prior to and following the stress task. Saliva is also collected at 10 and 20 minutes after the stress task. Heart rate will be measured through the duration of the stress task and recovery period.

The third visit includes a brief telephone call with the principal investigator to review participation in the study and answer any questions.

ELIGIBILITY:
Inclusion Criteria:

* Women ages 44-55 in the late perimenopause reproductive phase. Perimenopausal status will be determined based on menstrual cycle history. We will enroll women who have had an interval of amenorrhea of at least 60 days but <1 year consistent with the late menopause transition
* Participants in either group may be on antidepressant medications (for any indication), but doses must be stable within 30 days of study participation

Exclusion Criteria:

* History of bipolar diagnosis or primary psychotic disorder for both groups; prior history of depression in the no-perimenopausal depression group
* In the perimenopausal depression group, current depressive symptoms that are "severe" based on score of Center for Epidemiologic Studies Depression Scale (CES-D) >25.
* Current alcohol or substance use disorder
* Current suicidal ideation with intent and history of suicide attempt within 2 years of study participation
* Current or recent use of the following medications:

  1. Hormonal agents (e.g., hormone replacement therapy or combined oral contraceptive pills)within the past 30 days
  2. Oral, inhaled, or injected steroids within the past 90 days
  3. Blood pressure medications (e.g., Angiotensin-Converting Enzyme (ACE) inhibitors) within the past 90 days
  4. Antihistamines within the past two weeks
  5. Other medications determined by the study team to impact the RAAS (e.g., spironolactone).
* Current cigarette or nicotine use
* Current diagnosis of cardiovascular disease, type I or II diabetes, or other medical condition which the study team determines could impact study outcomes

Ages: 44 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-11-16 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Salivary aldosterone (pg/mL) levels at rest (before the stress task). | Immediately prior to the stress task.
  Examine variability in salivary aldosterone levels (pg/mL) by calculating medians.
Change in salivary aldosterone (pg/mL) levels in response to the stress task. | Immediately prior to the stress task and at intervals of 0, 10, and 20 minutes after the stress task.
  Examine variability in salivary aldosterone levels (pg/mL) in response to the TSST.
Plasma aldosterone (pg/mL) levels at rest (before the stress task). | Immediately prior to the stress task.
  Examine variability in plasma aldosterone levels (pg/mL) by calculating medians.
Change in plasma aldosterone (pg/mL) levels in response to the stress task. | Immediately prior to and at 0 minutes after the stress task.
  Examine variability in plasma aldosterone levels (pg/mL) in response to the TSST.
Plasma angiotensin II (pg/mL) levels at rest (before the stress task). | Immediately prior to the stress task.
  Examine variability in plasma angiotensin II levels (pg/mL) by calculating medians.
Change in plasma angiotensin II (pg/mL) levels in response to the stress task. | Immediately prior to and at 0 minutes after the stress task.
  Examine variability in plasma angiotensin II levels (pg/mL) in response to the TSST.
Plasma renin (pg/mL/hr) levels at rest (before the stress task). | Immediately prior to the stress task.
  Examine variability in plasma renin levels (pg/mL/hr) by calculating medians.
Change in plasma renin (pg/mL/hr) levels in response to the stress task | Immediately prior to and at 0 minutes after the stress task
  Examine variability in plasma renin levels (pg/mL/hr) in response to the TSST.

SECONDARY OUTCOMES:
Heart rate variability defined as the root mean square of successive differences (RMSSD) between normal heartbeats in ms values at rest (before the stress task). | Epoch recorded immediately before the stress task.
  Examine variability in RMSSD values measured at rest.
Change in heart rate variability defined as the root mean square of successive differences (RMSSD) between normal heartbeats in ms in response to the stress task. | Epochs recorded immediately before the stress task and intervals of 0, 10, and 20 minutes after the stress task.
  Examine variability in RMSSD values measured in response to the TSST.

CONTACTS AND LOCATIONS:
Overall Officials: Margo Nathan, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with the University of North Carolina.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: beginning at 9 and continuing for 36 months following publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.